CLINICAL TRIAL: NCT00249431
Title: A Pilot Study of Sertraline Plus Relapse Prevention Therapy (RP) for the Treatment of Pathological Gambling With Comorbid Abuse or Dependence
Brief Title: Effectiveness of Sertraline in Treating Pathological Gamblers With a Diagnosis of Alcohol Dependence - 1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to recruit patients.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #5156R; 5K23DA000482 (NIH)
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Alcoholism; Gambling
Keywords: Gambling; Alcohol
MeSH Terms: conditions — Alcoholism; Gambling | interventions — Sertraline; Secondary Prevention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Placebo and Relapse Prevention (Placebo Comparator): Patients will be treated with Relapse Prevention Therapy plus placebo
  Interventions: Behavioral: Relapse Prevention Therapy
- Sertraline and Relapse Prevention (Active Comparator): Patients will be treated with Relapse Prevention Therapy plus Sertraline.
  Interventions: Drug: Sertraline; Behavioral: Relapse Prevention Therapy

INTERVENTIONS:
Drug: Sertraline — Patients will be started on 25mg/day of Sertraline, and their dose will be increased to 50 mg/day by week two, and then weekly by 50mg/day based on clinical response and emergence of side effects. The maximum dose will be 200mg/day
  Other Names: zoloft
  Arms: Sertraline and Relapse Prevention
Behavioral: Relapse Prevention Therapy — Patients will have a weekly one-hour session for medication evaluation, relapse prevention therapy and answer questionnaires.

SUMMARY:
Pathological gamblers often are also dependent on alcohol and clinically depressed. Sertraline (Zoloft) is currently used to treat depression, panic disorder, and obsessive-compulsive disorder. The purpose of this trial is to determine the effectiveness of sertraline used in combination with relapse prevention therapy in decreasing gambling behavior and alcohol consumption in individuals with a diagnosis of pathological gambling and alcohol abuse or dependence.

DETAILED DESCRIPTION:
Alcohol abuse and depression commonly occur in conjunction with pathological gambling. Sertraline (Zoloft) is a selective serotonin reuptake inhibitor (SSRI) currently used to treat depression, panic disorder, and obsessive-compulsive disorder. The purpose of this trial is to determine the effectiveness of sertraline combined with relapse prevention therapy in decreasing gambling behavior and alcohol abuse.

Participants in this 10-week trial will be randomly assigned to receive either relapse prevention (RP) therapy and sertraline or RP therapy and a placebo. Participants will begin taking 25 mg of either sertraline or placebo in a single morning dose for one week. If, after one week, participants do not show improvement, the dose will increase to 50 mg per day during Week 2, and will increase by 50 mg per day every week thereafter to a maximal dose of 200 mg per day.

Weekly hour-long study visits will include a medication evaluation, RP therapy, and questionnaires. In addition, evaluations at baseline, Week 5, and Week 10 will include pathological gambling and depression ratings, urine drug screens, and biochemical measures of alcohol consumption and liver function. All other weekly study visits will include evaluation of side effects, an interview on alcohol use, measures related to obsessive-compulsive drinking, and assessments of vital signs and concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for pathological gambling
* Meets DSM-IV and SCID criteria for alcohol abuse or dependence
* Medically healthy

Exclusion Criteria:

* History of schizophrenia, schizoaffective disorder, or bipolar disorder
* Current diagnosis of substance abuse or dependence, other than alcohol or nicotine
* Current major depression
* Currently suicidal
* History of non-response to an adequate trial of sertraline, defined as 200 mg per day of sertraline for at least a 4-week period
* Previous treatment with relapse prevention therapy for pathological gambling or alcohol dependence within the 3 months prior to study entry
* Requires treatment with psychotropic medication
* Unwilling to consent to a drug-free period, according to the following: 2 weeks of abstinence from antidepressant drugs, other than fluoxetine, buspirone, lithium, anticonvulsants, barbiturates, opiates, or benzodiazepines; 4 weeks of abstinence from clonazepam; 5 weeks of abstinence from fluoxetine
* Clinically significant disorder, including kidney, pulmonary, cerebral vascular, cardiovascular, gastrointestinal, and endocrine disorders
* Abnormal laboratory tests
* Abnormal electrocardiogram
* Pregnant or breastfeeding
* Unwilling to use an adequate method of contraception for the duration of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2001-12 (Actual); Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Decreased gambling behavior; measured throughout study by the Clinical Global Impression Scale. | 10 weeks
  Decreased gambling behavior; measured throughout study by the Clinical Global Impression Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Blanco, M.D., Principal Investigator — Columbia University

REFERENCES:
- [Derived] Dowling N, Merkouris S, Lubman D, Thomas S, Bowden-Jones H, Cowlishaw S. Pharmacological interventions for the treatment of disordered and problem gambling. Cochrane Database Syst Rev. 2022 Sep 22;9(9):CD008936. doi: 10.1002/14651858.CD008936.pub2. PMID 36130734